CLINICAL TRIAL: NCT06070129
Title: Early Outcomes of Surgery in Patients With Massive and Sub Massive Pulmonary Embolism: ( a Single Center Experience)
Brief Title: Surgery in Pulmonary Embolisms
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohamed Emad Kamel, Assistant lecturer, Assiut University
Other Study IDs: surgery in pulmonary embolisms
Record Dates: First submitted 2023-09-30; First posted 2023-10-06 (Actual); Last update posted 2023-10-06 (Actual); Status verified 2023-09

CONDITIONS: Pulmonary Embolism
MeSH Terms: conditions — Pulmonary Embolism

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with massive pulmonary embolism or high-risk patients: * Characterized by evidence of low-cardiac-output syndrome or clinical shock attributed to PE as the underlying cause, based on 1 or more of the following: systemic arterial systolic blood pressure<90 mm Hg, need for positive inotrope or systemic vasoconstrictor support, need for mechanical circulatory support, cardiac arrest, or profound bradycardia (heart rate<40 bpm).
  * CT pulmonary angiography demonstrating a thrombus which occludes greater than 50% of the pulmonary artery (PA) cross-sectional area or occludes two or more lobar arteries.
  * Echocardiography both Trans thoracic and Trans esophageal shows right ventricular (RV) systolic dysfunction, RV dilation, or a RV/left ventricular (LV) diameter ratio of >0.9 on four chamber view.
  * Elevated cardiac troponin T and I above normal limits.
  Interventions: Procedure: surgical pulmonary embolectomy
- Patients with sub massive pulmonary embolism or intermediate -high risk: * Systolic blood pressure >90 mmHg and tachycardia (heart rate > 100 bpm).
  * CT pulmonary angiography shows that 30% to 50% of the pulmonary vasculature is occluded.
  * Echocardiography both Trans thoracic and Trans esophageal shows right ventricular (RV) systolic dysfunctions, RV dilation, or a RV/left ventricular (LV) diameter ratio of >0.9 on four chamber view.
  * Elevated cardiac troponin T and I above normal limits.
  Interventions: Procedure: surgical pulmonary embolectomy

INTERVENTIONS:
Procedure: surgical pulmonary embolectomy — open heart surgery with cardiopulmonary bypass with opening of the pulmonary artery and its major branches and extraction of the embolus

SUMMARY:
Measure early out comes of surgical pulmonary embolectomy in patients with massive and sub massive pulmonary embolism.

DETAILED DESCRIPTION:
* Pulmonary embolism (PE) is one of the most important causes of mortality in cardiovascular diseases. It represents the third cause of mortality after myocardial infarction and stroke.
* Risk factors of pulmonary embolism include malignancy, recent operation, hypercoagulability, and deep venous thrombosis (DVT). DVT is the most common risk factor.
* Acute pulmonary embolism is classified into massive or high risk (characterized by evidence of low-cardiac-output syndrome or clinical shock attributed to PE as the underlying cause, based on 1 or more of the following: systemic arterial systolic blood pressure<90 mm Hg, need for positive inotrope or systemic vasoconstrictor support, need for mechanical circulatory support, cardiac arrest, or profound bradycardia (heart rate<40 bpm)) and sub massive type or intermediate-high risk (characterized by evidence of adverse effects on the RV (dysfunction and strain), with mild hypotension, tachycardia, and 1 or more of the following: RV systolic hypo kinesis, RV dilatation by echocardiogram , elevated cardiac biomarkers (troponin I), elevated serum N-terminal pro brain natriuretic peptide, or electrocardiogram changes suggestive of RV strain.).
* Treatment options of acute massive and sub massive PE include systemic thrombolytic therapy, catheter directed thrombolysis (CDT) and surgical pulmonary embolectomy (SBE).
* The outcomes of the surgical treatment to the catheter-based treatment is still a topic of interest in management of acute pulmonary embolism.
* This study aims to measure early out comes of surgical pulmonary embolectomy in patients with massive and sub massive pulmonary embolism.

ELIGIBILITY:
Inclusion Criteria:

* Patient with massive pulmonary embolism or high-risk patients characterized by :

  * Evidence of low-cardiac-output syndrome or clinical shock attributed to PE as the underlying cause, based on 1 or more of the following: systemic arterial systolic blood pressure<90 mm Hg, need for positive inotrope or systemic vasoconstrictor support, need for mechanical circulatory support, cardiac arrest, or profound bradycardia (heart rate<40 bpm).
  * CT pulmonary angiography demonstrating a thrombus which occludes greater than 50% of the pulmonary artery (PA) cross-sectional area or occludes two or more lobar arteries.
  * Echocardiography both Trans thoracic and Trans esophageal shows right ventricular (RV) systolic dysfunction, RV dilation, or a RV/left ventricular (LV) diameter ratio of >0.9 on four chamber view.
  * Elevated cardiac troponin T and I above normal limits.

Patients with sub massive pulmonary embolism or intermediate -high risk characterized by:

* Systolic blood pressure >90 mmHg and tachycardia (heart rate > 100 bpm).
* CT pulmonary angiography shows that 30% to 50% of the pulmonary vasculature is occluded.
* Echocardiography both Trans thoracic and Trans esophageal shows right ventricular (RV) systolic dysfunction, RV dilation, or a RV/left ventricular (LV) diameter ratio of >0.9 on four chamber view.
* Elevated cardiac troponin T and I above normal limits

Exclusion Criteria:

* Patients less than 18 years of age.
* Low risk acute pulmonary embolism (less than 30% occlusion of pulmonary vasculature by CT pulmonary angiography, no signs of Rt ventricular systolic dysfunction, RV dilation or a RV/left ventricular (LV) diameter ratio of >0.9 on four chamber view by Echocardiography.
* Acute on top of chronic pulmonary embolism.

Min Age: 17 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: patients with massive and sub massive pulmonary embolism entering Assiut university hospital from October 2022 to November 2025 will be taken to be treated by surgical pulmonary embolectomy.
  patients will be divided according to type pulmonary embolism into two groups: massive pulmonary embolism group and sub massive pulmonary embolism group all of them will have the same inclusion and exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2023-11-01 (Estimated); Primary Completion 2025-11-01 (Estimated); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
mortality | baseline
  number of patients died
NYHA Functional Classification. | baseline
  I No limitation of physical activity. Ordinary physical activity does not cause undue fatigue, palpitation or shortness of breath.
  II Slight limitation of physical activity. Comfortable at rest. Ordinary physical activity results in fatigue, palpitation, shortness of breath or chest pain.
  III Marked limitation of physical activity. Comfortable at rest. Less than ordinary activity causes fatigue, palpitation, shortness of breath or chest pain.
  IV Symptoms of heart failure at rest. Any physical activity causes further discomfort.
right ventricular dimension | baseline
  dimensions of right ventricle in centimeter by echocardiography
left ventricular ejection fraction (EF %) | baseline
  left ventricular ejection fraction (EF ) percentage by echocardiography

SECONDARY OUTCOMES:
hospital stay days | baseline
  number of days the patient stayed at hospital after the surgery

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed EL-Minshawy, professor, Study Director — professor of cardiothoracic surgery surgery department; Sameh Abdelrahman, professor, Study Director — professor at cardiothoracic surgery department; Alaa Salah, lecturer, Study Director — lecturer at pulmonary disease department

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Goldberg JB, Spevack DM, Ahsan S, Rochlani Y, Dutta T, Ohira S, Kai M, Spielvogel D, Lansman S, Malekan R. Survival and Right Ventricular Function After Surgical Management of Acute Pulmonary Embolism. J Am Coll Cardiol. 2020 Aug 25;76(8):903-911. doi: 10.1016/j.jacc.2020.06.065. PMID 32819463
- [Background] Loyalka P, Ansari MZ, Cheema FH, Miller CC 3rd, Rajagopal S, Rajagopal K. Surgical pulmonary embolectomy and catheter-based therapies for acute pulmonary embolism: A contemporary systematic review. J Thorac Cardiovasc Surg. 2018 Dec;156(6):2155-2167. doi: 10.1016/j.jtcvs.2018.05.085. Epub 2018 Jun 8. PMID 30005883
- [Background] Meneveau N. Therapy for acute high-risk pulmonary embolism: thrombolytic therapy and embolectomy. Curr Opin Cardiol. 2010 Nov;25(6):560-7. doi: 10.1097/HCO.0b013e32833f02c5. PMID 20852415
- [Background] Azari A, Beheshti AT, Moravvej Z, Bigdelu L, Salehi M. Surgical embolectomy versus thrombolytic therapy in the management of acute massive pulmonary embolism: Short and long-term prognosis. Heart Lung. 2015 Jul-Aug;44(4):335-9. doi: 10.1016/j.hrtlng.2015.04.008. PMID 26077690
- [Background] Lin DS, Lin YS, Lee JK, Chen WJ. Short- and Long-Term Outcomes of Catheter-Directed Thrombolysis versus Pulmonary Artery Embolectomy in Pulmonary Embolism: A National Population-Based Study. J Endovasc Ther. 2022 Jun;29(3):409-419. doi: 10.1177/15266028211054763. Epub 2021 Oct 27. PMID 34706585
- [Background] Martinez Licha CR, McCurdy CM, Maldonado SM, Lee LS. Current Management of Acute Pulmonary Embolism. Ann Thorac Cardiovasc Surg. 2020 Apr 20;26(2):65-71. doi: 10.5761/atcs.ra.19-00158. Epub 2019 Oct 5. PMID 31588070